CLINICAL TRIAL: NCT00145769
Title: A Randomised Trial of Preoperative Radiotherapy for Stage T3 Adenocarcinoma of Rectum
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Gastro-Intestinal Trials Group (Network); Colorectal Surgical Society of Australasia (CSSA) (Unknown); Royal Australasian College of Surgeons (RACS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 01.04; NHMRC 209123 (Other Grant/Funding Number: National Health Medical and Research Council)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Adenocarcinoma of Rectum
Keywords: rectal cancer; radiotherapy; chemotherapy; chemoradiation; adjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Short Course Radiotherapy (Active Comparator): Short Course (SC) pre-operative radiotherapy, followed by surgery and adjuvant chemotherapy
  Interventions: Drug: Short Course Adjuvent Chemotherapy; Radiation: Short Course Radiotherapy
- Long Course Radiotherapy (Active Comparator): Long Course (LC) radiotherapy delivered with concurrent chemotherapy, followed by surgery and adjuvant chemotherapy
  Interventions: Drug: Long Course Adjuvant Chemotherapy; Radiation: Long Course Radiotherapy; Drug: Concurrent Chemotherapy
- Surgery (Active Comparator): Patients will receive initial surgery followed by post-operative management according to the NHMRC Guidelines for the prevention, early detection and management of colorectal cancer: Adjuvant therapy for rectal cancer.
  Interventions: Procedure: Initial Surgery

INTERVENTIONS:
Drug: Short Course Adjuvent Chemotherapy — Post operative adjuvant chemotherapy: 5FU (425mg/m2) preceded by Folinic acid (20mg/m2) delivered over 5 days for 6 monthly cycles
  Arms: Short Course Radiotherapy
Drug: Long Course Adjuvant Chemotherapy — Post operative adjuvant 5FU (425mg/m2) preceded by folinic acid (20mg/m2) delivered over 5 days for 4 monthly cycles
  Arms: Long Course Radiotherapy
Radiation: Short Course Radiotherapy — 25 Gy in 5 fractions over 5 days.
  Other Names: Radiation; RT; Short Course
  Arms: Short Course Radiotherapy
Radiation: Long Course Radiotherapy — 50.4 Gy delivered in 1.8 Gy fractions over 5 1/2 weeks.
  Other Names: Radiation; RT; Long Course
  Arms: Long Course Radiotherapy
Drug: Concurrent Chemotherapy — 5FU 225mg/m2/day delivered IV over continous 7 day period for the duration of radiotherapy (5 1/2 weeks).
  Arms: Long Course Radiotherapy
Procedure: Initial Surgery — Surgery is to be performed according to the NHMRC Guidelines for the prevention, early detection and management of colorectal cancer: Elective surgery for rectal cancer
  Arms: Surgery

SUMMARY:
This is a multi-centre randomised trial comparing long course (LC) preoperative chemoradiation with short course (SC) preoperative radiotherapy for patients with localised T3 rectal cancer.

DETAILED DESCRIPTION:
Objective:

* The objective is, in patients with T3 clinically resectable carcinoma of the rectum, to demonstrate that the local recurrence rate in patients treated with a long course (LC) of pre-operative radiotherapy with continuous infusion 5-FU is lower than that in patients treated with a short course (SC) of pre-operative radiotherapy with early surgery

Eligibility Criteria:

* The main eligibility criteria are that the patient has clinically resectable adenocarcinoma of the rectum, a clinical stage T3 tumour whose lower border is within 12 cm of the anal verge, and no evidence of distant metastases.

Endpoints:

* Primary endpoint is local recurrence.
* Secondary endpoints are overall survival, toxicity, abdminoperineal resection rate, quality of life.

Treatment arms:

* SC arm: Radiotherapy (RT) 25 Gy in 5 fr in 1 week to be followed by surgery within 1 week and 6 cycles of postoperative chemotherapy 5FU/Folinic acid.
* LC arm: RT 50.4 Gy in 28 fr in 5½weeks with 5FU 225 mg/m2/day throughout the course of RT, to be followed by surgery 4-6 weeks after completion of RT. 4 cycles of adjuvant 5FU/Folinic acid will be given.

ELIGIBILITY:
Inclusion Criteria:

All of the following must apply:

* Pathologically documented and clinically resectable adenocarcinoma of the rectum.
* The patient must be considered by the surgeon to be suitable for a curative resection.
* The patient must be considered by the radiation oncologist to have no contraindication to pre-operative radiotherapy.
* Clinical T3 stage tumour on endorectal ultrasound or MRI. When endorectal ultrasound cannot be performed satisfactorily due to a technical reason, such as stenosis or proximity of the tumour, and MRI is not available, infiltration of perirectal fat on CT scan is also acceptable.
* Tumour with lower border within 12 cm from anal verge on rigid sigmoidoscopy.
* ECOG performance status 0, 1 or 2.
* Adequate bone marrow function with neutrophil count at least 1.5 x 109/L and platelet count at least 100 x 109/L.
* Adequate liver function with bilirubin and alanine aminotransferase (ALT) <= 1.5 times the upper limit of normal.
* Adequate renal function with serum creatinine <= 1.5 times the upper limit of normal.
* Accessibility for treatment and follow-up.
* Written informed consent.

Exclusion Criteria:

* None of the following must apply:
* Evidence of distant metastases.
* Recurrent rectal cancer.
* Unstable cardiac disease or clinically significant active infection.
* Other cancer in the last 5 years except treated non-melanoma skin cancer or carcinoma in situ of the cervix.
* Pregnant or lactating females or female patients of childbearing potential who have not been surgically sterilized or are without adequate contraceptive measures.
* Contraindication to insertion of a suitable indwelling venous catheter e.g. implantable central venous device (infuse-a-port), Hickman catheter or peripherally inserted central catheter.
* Prior pelvic or abdominal radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2001-07; Primary Completion 2009-06 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Local recurrence | Main analysis will occur at minimum 3 years follow up of all patients. (After 6 years since start of trial)

SECONDARY OUTCOMES:
Survival | Main analysis will occur at minimum 3 years follow up of all patients. (After 6 years since start of trial)
Toxicity | Interim analyses will occur annually.
Abdominoperineal resection rate. This is defined as the proportion of all patients in any arm who undergo operation by abdominalperineal resection. | Main analysis will occur at minimum 3 years follow up of all patients. (After 6 years since start of trial)
Quality of life | Main analysis will occur at minimum 3 years follow up of all patients. (After 6 years since start of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ngan, FRANZCR, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (34):
- Australia (31):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Nepean Cancer Care Centre, Penrith, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Mater Private Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum Cancer Centre, Bendigo, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, East Bentleigh, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St Vincents Melbourne, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Andrew Love Cancer Centre, Geelong Hospital, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Murray Valley Private Hospital, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington

REFERENCES:
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Folkesson J, Birgisson H, Pahlman L, Cedermark B, Glimelius B, Gunnarsson U. Swedish Rectal Cancer Trial: long lasting benefits from radiotherapy on survival and local recurrence rate. J Clin Oncol. 2005 Aug 20;23(24):5644-50. doi: 10.1200/JCO.2005.08.144. PMID 16110023
- [Background] Ngan SY, Fisher R, Burmeister BH, Mackay J, Goldstein D, Kneebone A, Schache D, Joseph D, McKendrick J, Leong T, McClure B, Rischin D. Promising results of a cooperative group phase II trial of preoperative chemoradiation for locally advanced rectal cancer (TROG 9801). Dis Colon Rectum. 2005 Jul;48(7):1389-96. doi: 10.1007/s10350-005-0032-x. PMID 15906126
- [Derived] Ansari N, Solomon MJ, Fisher RJ, Mackay J, Burmeister B, Ackland S, Heriot A, Joseph D, McLachlan SA, McClure B, Ngan SY. Acute Adverse Events and Postoperative Complications in a Randomized Trial of Preoperative Short-course Radiotherapy Versus Long-course Chemoradiotherapy for T3 Adenocarcinoma of the Rectum: Trans-Tasman Radiation Oncology Group Trial (TROG 01.04). Ann Surg. 2017 May;265(5):882-888. doi: 10.1097/SLA.0000000000001987. PMID 27631775
- [Derived] Ngan SY, Burmeister B, Fisher RJ, Solomon M, Goldstein D, Joseph D, Ackland SP, Schache D, McClure B, McLachlan SA, McKendrick J, Leong T, Hartopeanu C, Zalcberg J, Mackay J. Randomized trial of short-course radiotherapy versus long-course chemoradiation comparing rates of local recurrence in patients with T3 rectal cancer: Trans-Tasman Radiation Oncology Group trial 01.04. J Clin Oncol. 2012 Nov 1;30(31):3827-33. doi: 10.1200/JCO.2012.42.9597. Epub 2012 Sep 24. PMID 23008301
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au